CLINICAL TRIAL: NCT03068936
Title: Intensity Modulated Radiotherapy Plus Cisplatin Versus Intensity Modulated Radiotherapy in Patients With Stage 2 Nasopharyngeal Carcinoma: A Phase 3 Multicenter, Open-label, Randomized, Non-inferior Clinical Trial
Brief Title: IMRT Plus Cisplatin Versus IMRT in Patients With Stage 2 Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1033400
Record Dates: First submitted 2017-02-15; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2016-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Intensity modulated radiotherapy; Cisplatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMRT group (Experimental): Intensity modulated radiotherapy once a day, 5 times a week, continuous treatment for about 6 weeks (DT 70Gy)
  Interventions: Radiation: Intensity modulated radiotherapy
- IMRT plus cisplatin group (Other): Intensity modulated radiotherapy once a day, 5 times a week, continuous treatment for about 6 weeks (DT 70Gy),plus synchronous cisplatin (100mg / m2 / times) chemotherapy, once every 3 weeks, a total of 2 times
  Interventions: Radiation: Intensity modulated radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy — Intensity modulated radiotherapy once a day, 5 times a week, continuous treatment for about 6 weeks (DT 70Gy)
  Other Names: IMRT
Drug: Cisplatin — Synchronous cisplatin (100mg / m2 / times) chemotherapy, once every 3 weeks, a total of 2 times
  Arms: IMRT plus cisplatin group

SUMMARY:
Nasopharyngeal carcinoma has high incidence in the southern China, especially in Guangdong Province. In the world, the standardized morbidity has reached 30/10 million in men while in women, about 13/10 million. At present, the incidence of nasopharyngeal carcinoma in China accounted for more than 80% of the world. The cancer-related deaths is in the eighth, which is a serious threat to our people's health and life. A recent multi-center phase II study of stage II nasopharyngeal carcinoma showed that: compared with Intensity Modulation Radiotherapy (IMRT) plus cisplatin, the 3 year local control rate, regional control rate, distant metastasis-free survival rate and disease-specific survival rate of IMRT were similar, but the side effects of radiotherapy alone group were lower.

Based on the results of the phase II clinical study, the investigators designed this phase III clinical study, with the aim to compared the efficacy and toxicity of these two treatment programs. And finally to provide sufficient evidence for the treatment of stage II nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* The sex of the subject is not limited, the age is from 18 to 70 years old;
* Histologically proven nasopharyngeal squamous cell carcinoma, World Health Organization (WHO) II-III type;
* Union Internationale Contre le Cancer(UICC) stage 9 clinical stage II patients；
* Karnofsky score ≥ 80 points;
* No evidence of distant metastasis;
* Having an nasopharyngeal MRI before treatment ,which can measure the size of the tumor in order to analyze the effect.

Exclusion Criteria:

* The subject had previously suffered from other malignancies (except non-melanotic skin cancer or cervical carcinoma in situ);
* Previously received immunotherapy;
* Previously received chemotherapy;
* Previously received radiation therapy;
* Patients who had previously undergone surgical treatment for head and neck tumors (excluding cervical lymphadenectomy);
* Evidence of distant metastases or other malignancies at the same time.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | up to 3 years
  Refers to the time from included to death due to any cause.

IPD SHARING:
Plan to Share IPD: No